CLINICAL TRIAL: NCT03301519
Title: Genetics of Beta Cell Failure in Mexican Americans
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Thomas Buchanan, Professor of Medicine, University of Southern California
Other Study IDs: HS 013025
Record Dates: First submitted 2017-09-21; First posted 2017-10-04 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Gestational Diabetes; Diabetes Type 2; Insulin Resistance; Beta Cell Function; Genetics; Nutrition; Physical Activity; Adipokines; Obesity; Air Pollution
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2; Insulin Resistance; Motor Activity; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, plasma samples from oral glucose tolerance test, plasma samples from intravenous glucose tolerance test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a family based genotype-phenotype study designed to assess genetic and environmental influences on obesity, insulin resistance and beta cell function in the context of gestational diabetes.

DETAILED DESCRIPTION:
Mexican American women with prior gestational diabetes and their first degree relatives and Mexican American women with prior normal glucose tolerance in pregnancy are studied with detailed phenotyping consisting of oral and intravenous glucose tolerance tests, body composition studies, diet and physical activity assessments, and circulating biomarkers potentially related to obesity, insulin resistance, pancreatic beta cell function, gestational diabetes and type 2 diabetes. Spouses of the gestational diabetic and control probands are studied with oral glucose tolerance tests. Offspring of the gestational and control probands have fasting glucose determinations. All participants provide DNA for genetics testing. A subset of the gestational diabetic probands and their first degree relatives return 3-5 years after baseline testing for repeat phenotyping.

ELIGIBILITY:
INCLUSION CRITERIA

1. Probands with Prior Gestational Diabetes Mellitus ("GDM PROBANDS")

   * Mexican American (parents and at least 3/4 four grandparents
   * age >18 years
   * GDM in singleton pregnancy in prior 5 years
   * impaired glucose levels or sum of five OGTT glucose values >625 mg/dl on 75 gram oral glucose tolerance test
   * Fasting plasma glucose <126 mg/dl
   * At least two adult siblings of cousin not known to have diabetes and available for phenotyping; .
2. Siblings and Cousins of GDM Probands

   * Full sibling or first cousin of GDM proband
   * Age >18 yrs
   * Fasting plasma glucose <126 mg/dl.
3. Parents, Uncles and Aunts of GDM Probands

   * Full blooded parent, uncle or aunt of GDM proband
4. Control Proband

   * Mexican American as defined for GDM probands
   * One glucose challenge test result <120 mg/dl at >24 weeks gestation
   * No diabetes in first degree relative
   * Frequency matched to GDM probands by distributions of age, BMI and parity.
5. Spouse of GDM or Control Proband

   * Spouse of GDM proband
   * Age >18
   * At least one child with proband able to provide DNA
6. Child of Proband

   * Child of GDM or control proband and spouse who provided DNA

EXCLUSION CRITERIA

1. PROBANDS (GDM OR CONTROL):

   * Chronic medical illness or medication known to alter glucose/insulin metabolism
   * Current pregnancy or breastfeeding
   * Ilicit drug or alcohol abuse,
   * Inability or unwillingness to give informed consent.
2. SIBLINGS AND COUSINS OF PROBANDS:

   * Chronic medical illness or medication known to affect glucose/insulin metabolism
   * Current pregnancy or breastfeeding,
   * Ilicit drug or alcohol abuse
   * Inability or unwillingness to give informed consent.
3. PARENTS OF PROBANDS

   * Inability or unwillingness to give informed consent.
4. SPOUSE OF GDM or CONTROL PROBAND

   * Inability or unwillingness to give informed consent.
5. CHILD OF GDM or CONTROL PROBAND

   * Lack of parent consent or child assent.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: See Inclusion and Exclusion Criteria
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Actual)
Dates: Start 2001-07-01 (Actual); Primary Completion 2013-05-31 (Actual); Study Completion 2013-05-31 (Actual)

PRIMARY OUTCOMES:
Pancreatic Beta Cell Compensation for Insulin Resistance | Single time point for primary cohort, repeated 4.5 years later in subset
  Disposition index from intravenous glucose tolerance test

SECONDARY OUTCOMES:
Insulin Senstivity | Single time point for primary cohort, repeated 4.5 years later in subset
  Si from computer modeled intravenous glucose tolerance test
Acute Insulin Release | Single time point for primary cohort, repeated 4.5 years later in subset
  Incremental area under insulin curve during first 10 minutes intravenous glucose tolerance test
Glucose tolerance | Single time point for primary cohort, repeated 4.5 years later in subset
  normal, impaired or diabetic glucose level determined using American Diabetes Associate criteria applied to glucose levels from a 2-hour, 75 gram oral glucose tolerance test
Diabetes type 2 | Single time point for primary cohort, repeated 4.5 years later in subset
  Fasting glucose >125 mg/dl and/or 2-hour glucose on 75 gram oral glucose tolerance test >199 mg/dl
Dietary Intake | Single time point for primary cohort, repeated 4.5 years later in subset
  Measured by semi-quantitative Harvard Food Frequency Questionnaire
Physical Activity | Single time point for primary cohort, repeated 4.5 years later in subset
  Measured by Multi-ethnic Cohort Physical Activity Questionnaire
Body Fat | Single time point for primary cohort, repeated 4.5 years later in subset
  Percent body fat measured by dual photon X-ray absorptiometry
Circulating adipokine levels | Single time point for primary cohort, repeated 4.5 years later in subset
  Fasting levels of approximately 20 adipocytokines

IPD SHARING:
Plan to Share IPD: No